## Single Session Pain Catastrophizing Class: Efficacy & Mechanisms for Reducing Opioid Use Among Chronic Pain Patients

Statistical Analysis Plan NCT03950791 4/1/2024

## **Statistical Analysis Plan**

To test the hypothesis that the Empowered Relief class would lead to greater reductions in opioid use than Health Education class, the primary outcome/endpoint was designated as reduction in opioid use as represented by morphine equivalent dose (MED) at 3 months. Within-participant differences from baseline to 3 months in MED was calculated. As the MED scores and difference scores were not normally distributed, the comparison between difference scores in the Empowered Relief arm and the Health Education arm utilized a Mann-Whitney U test (primary outcome).

We then compared the proportion of participants reaching clinically significant reductions in MED between the Empowered Relief and Health Education groups. Clinically minimal reduction is defined as >15% reduction in opioid use. We quantified absolute opioid reduction in addition to percent change reduction within subject and between groups. Finally, we quantified percent achieving each group threshold for importance of change (15%, 30%, and 50% as minimally, moderately, and substantially important change scores, respectively).